CLINICAL TRIAL: NCT01247909
Title: An Open Randomised Trial of Ceftriaxone v Penicillin and Gentamicin in Infant Severe Sepsis and Bacterial Meningitis in Malawi
Brief Title: Infant Severe Sepsis and Bacterial Meningitis in Malawi
Acronym: Infaseme
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Elizabeth Molyneux, Professor of Paediatircs, Kamuzu University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Infaseme
Record Dates: First submitted 2010-01-14; First posted 2010-11-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Infant Bacterial Meningitis
MeSH Terms: interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftriaxone (Experimental): Ceftriaxone in infants with sepsis and bacterial meningitis
  Interventions: Drug: Ceftriaxone v penicillin and gentamicin
- Penicillin and gentamicin (Active Comparator): Penicillin and Gentamicin in infants with sepsis and bacterial meningitis
  Interventions: Drug: Ceftriaxone v penicillin and gentamicin

INTERVENTIONS:
Drug: Ceftriaxone v penicillin and gentamicin — Ceftriaxone v the standard treatment of infant meningitis (penicillin and gentamicin). Ceftriaxone will be given at a dose of 80mg/kg once a day for at least 14 days.

SUMMARY:
This study aims to improve the outcome of infants (<2 months) with severe sepsis and meningitis at the Queen Elizabeth Central Hospital, Blantyre, Malawi.

Currently WHO recommends the treatment of infant severe sepsis and bacterial meningitis with 14 to 21 day course of penicillin and gentamicin as first line. The second line treatment is cefotaxime or ceftriaxone.

Severe bacterial infections are common in infants under 2 months of age and the mortality is very high (~50%). There are several reasons for this; one is that the first line antibiotics used are no longer as effective as they used to be. Bacterial resistance to the first line antibiotics has increased and some infections especially of the central nervous system may only be partly treated and not eradicated by present therapy. First line treatment is cheap and available but requires 4 injections a day, for at least 14 days, a total of 58 injections. Many mothers find this number too much and abscond. The investigators second line therapy is ceftriaxone which is also available and cheap and the advantage of being given as a daily injection. The disadvantage is that it can cause (reversible) jaundice particularly in premature babies and it must not be given with calcium products. The investigators do not give calcium to the investigators infants as the investigators cannot routinely check electrolytes. All the most common causes of bacterial meningitis in this age group in the investigators setting are sensitive to ceftriaxone.

The investigators wish to undertake an open randomized trial of penicillin and gentamicin v ceftriaxone as first line treatment for infant meningitis. The investigators are able to monitor for side effects.

The investigators hypothesise that the ceftriaxone arm will have 20% less deaths that the penicillin and gentamicin group.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 2 months
* Suspicion of bacterial meningitis
* Parental/guardian informed consent

Exclusion Criteria:

* Infant with hyperbilirubinaemia
* Infant requiring calcium
* Infant know to be hypersensitive to any of the three drugs
* Infant who has been an inpatient for more than 72 hours
* Infant with congenital central nervous system abnormalities

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 351 (Actual)
Dates: Start 2010-04; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Recovery v death or severe residual neurological sequelae at hospital discharge, 1 month and 6 months post discharge. | 3 years

SECONDARY OUTCOMES:
Outcome by causative bacterial agent, recovery v death or severe residual neurological sequelae at hospital discharge, 1 month and 6 months post discharge. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Molyneux, FRCPCH, Principal Investigator — Malawi College of Medicine, Paediatrics Department
Locations (1):
- Queen Elizabeth Central Hospital/ College of Medicne, Private Bag 360 Blantyre, Malawi